CLINICAL TRIAL: NCT00499304
Title: Diagnosing Expiratory Flow Limitation in COPD Patients With the Forced Oscillation Technique Using Linear Regression in the Time Frequency Domain
Brief Title: Forced Oscillation Technique (FOT) and Expiratory Flow Limitation (EFL)
Status: Completed | Type: Observational
Sponsor: Medical Center Alkmaar (Other)
Other Study IDs: NL13873.09406
Record Dates: First submitted 2007-07-10; First posted 2007-07-11 (Estimated); Last update posted 2008-06-06 (Estimated); Status verified 2008-06

CONDITIONS: COPD
Keywords: Forced oscillation Technique (FOT); Expiratory flow limitation (EFL); Breathing artifacts; COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of this study is to distinguish COPD patients with expiratory flow limitation in body plethysmography (open loop) from the patients without expiratory flow limitation in body plethysmography (closed loop) with the obtained FOT parameters.

DETAILED DESCRIPTION:
In daily practice the expiratory flow limitation is measured by body plethysmography. An open loop in body plethysmography shows expiratory flow limitation in COPD patients. But body plethysmography requires that the patient quietly sits in a closed box and is not able to follow changes breath by breath. The goal of this study is to validate the Forced oscillation technique (FOT) for measuring expiratory flow limitation in COPD patients.30 COPD patients with an open loop in body plethysmography are compared to 30 COPD patients with a closed loop. The methods used in this study are the maximal overlap discrete short time Fourier transform (MODFT) combined with a total least squares analysis. It is hypothesized that the obtained FOT parameters are able to distinguish the patients with expiratory flow limitation in body plethysmography from the patients without expiratory flow limitation in body plethysmography.Secondary study questions are: 1) to what extend are the FOT parameters distorted by breathing artifacts and measurement noise. 2)What changes can be detected by FOT in expiratory flow limitation after administration of salbutamol.

ELIGIBILITY:
Inclusion Criteria:

* Presenting to the outpatient clinic
* Age 50-80 years
* Diagnosed with COPD according to the standard criteria
* Gold Stage II to IV COPD
* Current or ex-smokers (at least 10 PY)
* Stable disease (No current exacerbation or exacerbation during the 4 weeks previous to the inclusion)

Exclusion Criteria:

* History of exacerbation of COPD in the preceding month
* Upper airway obstruction
* Allergic Asthma
* OSAS (obstructive sleep apnea syndrome)
* Extreme obesity (BMI>35)
* Clinically manifest cardiac disease (for example clinically relevant congestive heart failure, unstable angina pectoris)

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Stable GOLD 2-4 COPD patients
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2006-11; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dewi Tjiong, drs, Principal Investigator — Medical Center Alkmaar
Locations (1):
- Medical Center Alkmaar, Alkmaar, Netherlands